CLINICAL TRIAL: NCT02113202
Title: Visualization of a VEGF-targeted Near-Infrared Fluorescent Tracer in Patients With Familial Adenomatous Polyposis During Fluorescence Endoscopy A Single Center Pilot Intervention Study
Brief Title: Molecular Fluorescence Endoscopy in Patients With Familial Adenomatous Polyposis, Using Bevacizumab-IRDye800CW
Acronym: FLUOFAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL45148.042.13; 2013-002490-22 (EudraCT Number)
Record Dates: First submitted 2014-04-02; First posted 2014-04-14 (Estimated); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Adenomatous Polyposis Coli
Keywords: Optical imaging; Fluorescence endoscopy; Near infrared fluorescence; Familial Adenomatous Polyposis; IRDye800CW; Vascular Endothelial Growth Factor A; Gastrointestinal endoscopy
MeSH Terms: conditions — Adenomatous Polyposis Coli

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tracer dose: 4.5 mg (Experimental): Patients receive three days before the fluorescence endoscopy procedure (with the near infrared fluorescence endoscopy platform) 4.5 mg of the fluorescent tracer bevacizumab-IRDye800CW.
  Interventions: Drug: Bevacizumab-IRDye800CW; Device: Near infrared fluorescence endoscopy platform
- Tracer dose: 10 mg (Experimental): Patients receive three days before the fluorescence endoscopy procedure (with the near infrared fluorescence endoscopy platform) 10 mg of the fluorescent tracer bevacizumab-IRDye800CW.
  Interventions: Drug: Bevacizumab-IRDye800CW; Device: Near infrared fluorescence endoscopy platform
- Tracer dose: 25 mg (Experimental): Patients receive three days before the fluorescence endoscopy procedure (with the near infrared fluorescence endoscopy platform) 25 mg of the fluorescent tracer bevacizumab-IRDye800CW.
  Interventions: Drug: Bevacizumab-IRDye800CW; Device: Near infrared fluorescence endoscopy platform

INTERVENTIONS:
Drug: Bevacizumab-IRDye800CW — Intravenous administration of a 4.5 mg, 10 mg or 25 mg of Bevacizumab-IRDye800CW 3 days prior to the fluorescence endoscopy procedure.
  Other Names: Beva-800CW; Bevacizumab-800CW; Avastin-800CW (Roche)
Device: Near infrared fluorescence endoscopy platform — A flexible fiber-bundle is attached with its proximal end to a camera which can detect near infrared fluorescent light. The distal end is inserted into the working channel of a clinical video endoscope, which is used for the surveillance endoscopy procedure.

SUMMARY:
There is a need for better visualization of polyps during surveillance endoscopy in patients with hereditary colon cancer syndromes like Familial Adenomatous Polyposis (FAP) and Lynch Syndrome (LS), to improve the adenoma detection rate. Optical molecular imaging of adenoma associated biomarkers is a promising technique to accommodate this need. The biomarker Vascular Endothelial Growth Factor (VEGF) is overexpressed in adenomatous colon tissue versus normal tissue and has proven to be a valid target for molecular imaging. The University Medical Center Groningen (UMCG) developed a fluorescent tracer by labeling the VEGF-targeting humanized monoclonal antibody bevacizumab, currently used in anti-cancer therapy, with the fluorescent dye IRDye800CW. The investigators hypothesize that when bevacizumab-IRDye800CW is administered to patients, it accumulates in VEGF expressing adenomas, enabling adenoma visualization using a newly developed near-infrared (NIR) fluorescence endoscopy platform (NL43407.042.13). This hypothesis will be tested in this feasibility study, next to the determination of the optimal tracer dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients with genetically or clinically proven Familial Adenomatous Polyposis. Genetically proven: Adenomatous Polyposis Coli (APC)-mutation identified. Clinically proven: more than 100 colorectal polyps at diagnosis
* Age 18 to 70 years
* Written informed consent
* Adequate potential for follow-up

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent
* Proctocolectomy
* MutYH mutation
* Concurrent uncontrolled medical conditions
* Pregnant or lactating women. Documentation of a negative pregnancy test must be available for woman of childbearing potential. Woman of childbearing potential are pre-menopausal women with intact reproductive organs and women less than two years after menopause.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of fluorescent adenomatous polyps during surveillance endoscopy using the near-infrared fluorescence endoscopy platform in patients with Familial Adenomatous Polyposis (FAP), after administration of the fluorescent tracer bevacizumab-IRDye800CW. | At surveillance endoscopy
  The main objective of this study is to determine the sensitivity of the fluorescent tracer bevacizumab-IRDye800CW and the near-infrared fluorescence endoscopy platform in identifying adenomatous polyps during surveillance endoscopy in patients with Familial Adenomatous Polyposis (FAP).

SECONDARY OUTCOMES:
Meassure the mean fluorescent intensity of the polyps during fluorescence endoscopy, resect the polyps and score VEGF intensity after immunohistochemistry for VEGF. | Two years
  In this outcome meassure, it is determined if there is a correlation between the observed mean fluorescence intensity of a polyp and the VEGF expression in the same polyp, as determined with immunohistochemistry and eventually RNA/DNA analysis. In other words, does the mean fluorescence intensity reflect the VEGF expression of the polyp?
Number of participants with Serious Adverse Events as a measure of safety and Tolerability. | Up to 1 week after administration
  Collection of safety data regarding administration of Bevacizumab-IRDye800CW (adverse events (AE), serious adverse events (SAE) and suspected unexpected serious adverse reactions (SUSAR)).
Measure the mean fluorescent intensity of adenomas and compare this between the three different dosing groups to determine the best tracer dose for the fluorescence endoscopy procedure. | Two years
  The goal of this outcome measure, is to determine the optimal tracer dose (4.5, 10 or 25 mg) of bevacizumab-IRDye800CW for the molecular-guided fluorescence endoscopy procedure to visualize adenomas. The fluorescence intensity of adenomas will be measured in vivo during fluorescence endoscopy and ex vivo (e.g. using confocal fluorescence microscopy, spectroscopy). This will be compared between the three subgroups (patients with different time intervals between tracer injection and endoscopy procedure) to determine the best time interval between tracer injection and endoscopy procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Wouter B Nagengast, PharmD MD PhD, Principal Investigator — University Medical Center Groningen; Jan Jakob Koornstra, MD PhD, Principal Investigator — University Medical Center Groningen; Jan H Kleibeuker, MD, senior full professor, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands